CLINICAL TRIAL: NCT06309875
Title: Effect of the PLAN CUIDARTE on the Caregiving Competence of People With Heart Failure: Implementation of the Research Protocol.
Brief Title: Effect of the PLAN CUIDARTE on the Caregiving Competence of People With Heart Failure
Acronym: PLANCUIDARTE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad de la Sabana (Other)
Collaborators: Universidad de Caldas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENF- 25-2018
Record Dates: First submitted 2024-02-20; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Caregiver Burden; Discharge Plan; Care Transitions; Nursing
MeSH Terms: conditions — Heart Failure; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: A pre-post test Randomized Clinical Trial (RCT) is proposed with a comparison group, with blinding of the participants with blinding of the participants, with application of a pilot test beforehand. pilot test.
  The intervention group is established as the group that receives the PLAN CUIDARTE (intervention described later) and as a comparison group the one receiving the conventional discharge plan (described later)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Set of specific activities carried out by the health care team by the health care team at the time of hospital discharge of HF patients: the patients with HF:
  Interventions: Other: Conventional care
- PLAN CUIDARTE (Experimental): The "PLAN CUIDARTE" is an intervention aimed at addressing the hospital discharge of people with HF, based on the nursing theory of transitions of Afaf Meleis(46) and under the guidelines of Robin Whittemore for the systematic development of complex interventions for experimental type research in nursing. The PLAN CUIDARTE addresses the specific educational needs of HF patients, as established by the patients with HF, as established by international accreditation standards.
  Interventions: Other: PLAN CUIDARTE

INTERVENTIONS:
Other: PLAN CUIDARTE — Description Plan Cuidarte
  Arms: PLAN CUIDARTE
Other: Conventional care — Description Conventional care
  Arms: Conventional

SUMMARY:
According to the World Health Organization (WHO), by 2021 cardiovascular diseases (CVD) will be a public health problem, among them heart failure (HF), since this is a chronic disease, patients should be competent in their care. Despite the above, according to research conducted in Colombia, 59.7% of people with chronic noncommunicable diseases (NCDs) have a level of care competence considered not optimal; patients report not having sufficient knowledge of the disease or experience feelings of lack of tools for the management of symptoms and the challenges of post-hospitalization.

The objective of the research is to determine the effect of the PLAN CUIDARTE on the caregiving competence of people with HF

Methodology: Pre-posttest randomized clinical trial, with blinding of the participants, where the intervention "PLAN CUIDARTE" is applied and the initial and subsequent caregiving competence is evaluated in the comparison group and in the intervention group for pretest - posttest and between-group comparisons.

DETAILED DESCRIPTION:
Eligibility Criteria:

Inclusion criteria

* Patients over 18 years of age with a diagnosis of HF.
* Patients with HF who are hemodynamically stable.
* Patients with SPMSQ - PFERFFER of 0 - 4 errors or 5 errors, patient who has not received primary education.
* Patient with a PULSES of 6 to 11

Exclusion criteria

* Patients with heart failure with heart transplantation scheduled in the next 6 months.
* Patients requiring transfer to an intensive or intermediate care unit.

Outcome Measures:

* Primary: Caring competence.
* Secondary: Satisfaction with care

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who are hospitalized and admitted to the institution with a diagnosis of HF decompensation with a time of diagnosis greater than 6 months.
* Patients who are hemodynamically stable, without alteration of the state of consciousness.

Exclusion Criteria:

* HF patients who are hospitalized for cardiac transplantation,
* Who are under palliative management or who, at the time of discharge, have a formal
* Who have a designated formal caregiver or are discharged to an institution other than home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-11-12 (Estimated)

PRIMARY OUTCOMES:
Care Competence | 30 days
  capacity, ability and preparation of the patient or family caregiver to the patient or family caregiver to perform the task of caregiving(4), which is made up of the following five dimensions: knowledge five dimensions: knowledge, uniqueness, instrumental, enjoyment, anticipation and social relationship, uniqueness, instrumental, enjoyment, anticipation and social relationship.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Caldas, Manizales, Caldas Department, Colombia

IPD SHARING:
Plan to Share IPD: No